CLINICAL TRIAL: NCT06155721
Title: Desarrollo y evaluación de Experiencias en Realidad Virtual Para la estimulación Cognitiva en el Centro Sociosanitario El Carme de Badalona Servicios Asistenciales (BSA)
Brief Title: Development and Evaluation of Virtual Reality Experiences for Cognitive Stimulation at the Sociosanitary Center El Carme
Acronym: RTCSSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badalona Serveis Assistencials (Other)
Collaborators: Public Health Agency of Barcelona (Other); Reality Telling SL (Unknown)
Responsible Party: Principal Investigator, Jose Ferrer Costa, Principal Investigator, Badalona Serveis Assistencials
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PI-23-195
Record Dates: First submitted 2023-11-03; First posted 2023-12-04 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Dysfunction; Mild Cognitive Impairment
Keywords: Cognitive Stimulation; Virtual Reality; Mild Cognitive Impairment; Cognitive Rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a single-arm interventional study where all participants receive the same intervention- a cognitive stimulation program administered through virtual reality (VR). Participants with mild to moderate cognitive impairment will engage in structured VR sessions aimed at stimulating cognitive functions, particularly attention and memory. The study will monitor participants' cognitive performance through standardized cognitive scales pre- and post-intervention, as well as gather subjective feedback on their experience to evaluate acceptability and motivation. Additionally, healthcare professionals' perceptions of the VR intervention's applicability to clinical practice will be assessed through structured interviews or questionnaires.
Masking Description: No masking was involved in this study as all participants received the same intervention (the cognitive stimulation program using virtual reality created in collaboration with Reality Telling SL), and the open-label nature of the intervention made it impractical to blind participants or researchers to the treatment being provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Cognitive Stimulation Program (Experimental): Participants with MCI undergo 8 VR sessions, using Oculus Quest 2 headsets for immersive cognitive exercises. Activities include a Supermarket Shopping Task for memory, a Payment Task for cognitive flexibility, and a Recipe Sequencing Task for problem-solving. Additionally, 360-degree videos with visuo-verbal stimulation are used to engage attention and episodic memory, monitored by therapists.
  The investigators employ Oculus Quest 2 VR headsets with hand tracking technology to provide a seamless and immersive experience, especially beneficial for participants with Mild Cognitive Impairment (MCI).
  Interventions: Device: Virtual Reality Cognitive Stimulation Program

INTERVENTIONS:
Device: Virtual Reality Cognitive Stimulation Program — Intervention Type: Device Intervention Name: Virtual Reality Cognitive Stimulation Program Description: This program utilizes virtual reality to conduct cognitive stimulation exercises aimed at improving memory, executive functions, and attention in individuals with Mild Cognitive Impairment (MCI). It includes interactive tasks such as virtual shopping, payment simulations, and recipe sequencing, along with 360-degree video sessions for attention and episodic memory training.

SUMMARY:
The goal of this clinical trial is to test a virtual reality (VR)-based program designed for cognitive stimulation in individuals attending the conventional cognitive rehabilitation program at the Day Hospital of CSSC (Centro Sociosanitario El Carme) in Badalona, Spain. The trial will specifically assess VR's impact on declarative memory and executive functions through interactive exercises, as well as attention and episodic memory through VR video stimuli.

The main questions it aims to answer are:

* Will patients with mild cognitive impairment find the VR program enjoyable and easy to use?
* Can VR interventions help improve patients' cognitive functions, specifically attention and memory?
* Do healthcare professionals find VR a practical tool for cognitive stimulation in their clinical practice?

Participants will undergo a series of 8 sessions, scheduled twice a week to coincide with the conventional rehabilitation appointments. The VR equipment used will be Oculus Quest 2 headsets, offering an immersive experience with hand-tracking technology that simplifies interactions, particularly beneficial for those with mild cognitive impairment (MCI). During the study, participants will:

* Engage with a VR-based cognitive stimulation program.
* Undergo assessments of the participants´ cognitive functions before and after the intervention.
* Provide feedback on the participants´ experience with the VR program.

Researchers will analyze the data to see if:

* The VR program leads to noticeable improvements in the cognitive abilities of participants.
* The program is well-received and deemed beneficial by both patients and healthcare professionals.

DETAILED DESCRIPTION:
Background:

Cognitive impairment affects a significant portion of the aging population, leading to challenges in daily functioning and a reduced quality of life. Traditional cognitive rehabilitation techniques have shown benefits, but patient engagement and adherence remain challenging. Innovations such as virtual reality (VR) offer new avenues for cognitive stimulation, potentially enhancing patient involvement and treatment outcomes.

Study Design:

This clinical trial aims to evaluate the acceptability and efficacy of a VR-based cognitive stimulation program among patients with mild to moderate cognitive impairment at Centro Sociosanitario El Carme in Badalona. It will employ a pretest-posttest design to assess cognitive changes, utilizing standardized cognitive scales and gathering qualitative feedback on user experience.

Objectives:

Primary Objective: To assess the acceptability of the VR-based cognitive stimulation program among patients with mild to moderate cognitive impairment.

Secondary Objectives:

To evaluate whether the VR interventions are perceived as engaging and motivating by the patients, which would suggest positive adherence to the cognitive stimulation program.

To measure changes in cognitive performance, particularly in attention and memory, pre- and post-intervention, to determine the effectiveness of the program.

To understand healthcare professionals' perceptions of the applicability of VR interventions in clinical practice for cognitive stimulation.

To identify potential improvements for the implementation of the VR program based on patient and healthcare staff feedback.

To gather data that could be useful for the development of future VR experiences aimed at patients with cognitive impairments.

Methodology:

Participants will be recruited from the Centro Sociosanitario El Carme and will undergo an initial assessment to establish a cognitive baseline. The participants will then engage in a series of VR sessions designed to provide cognitive stimulation. The program will focus on exercises to enhance attention and memory, incorporating interactive elements to maintain engagement. After completing the sessions, participants will be re-assessed using the same cognitive scales.

Feedback on the VR experience will be collected through structured interviews and questionnaires to gauge acceptability, perceived usefulness, and motivation. Healthcare professionals involved in the administration of the VR program will also be interviewed to understand their views on the integration of VR into therapeutic practices.

Expected Outcomes:

It is hypothesized that the VR program will be well-received by patients, evidenced by high rates of program completion and positive subjective feedback. Post-intervention improvements in cognitive scale scores are expected, indicating the potential efficacy of VR-based stimulation. Insights from healthcare professionals are anticipated to highlight the practicality of VR in clinical settings and suggest improvements for future applications.

Relevance:

The findings from this trial could support the adoption of VR technologies in cognitive rehabilitation, offering a novel, scalable, and potentially more effective approach to managing cognitive impairments. The study may also contribute to the evidence base required for integrating technological innovations into standard healthcare practice.

Conclusion:

By exploring the intersection of VR technology and cognitive rehabilitation, this study seeks to advance the understanding of innovative treatments for cognitive impairments and foster improved patient outcomes through enhanced engagement and stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be classified as having mild cognitive impairment with a Mini-Mental State Examination (MMSE) score greater than 23.
* Participants must be currently attending cognitive rehabilitation sessions at the Day Hospital of the Centro Sociosanitario El Carme (CSSC).
* Participants must be able to give informed consent or, in the case of incapacity, consent must be obtained from their legal representative.

Exclusion Criteria:

* Patients with a severe or unstable illness that could interfere with participation in the study.
* Patients with serious psychiatric disorders, such as psychotic disorders, delusions, or hallucinations that may be exacerbated by the use of virtual reality.
* Patients with severe visual limitations that would prevent the use of virtual reality.
* Presence of ocular diseases causing blurred vision that cannot be corrected with contact lenses or glasses.
* Presence of auditory pathologies that cause a significant decrease in hearing without hearing aids.
* High sensitivity to motion sickness.
* Subjects with epilepsy.
* Patients who are unable or unwilling to give informed consent.

Withdrawal Criteria

The emergence of health problems that could interfere with the continuity of participation in the study, or the withdrawal of consent by the participant.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Ferrer Costa, MD, Principal Investigator — Medical Researcher and Project Manager
Locations (1):
- Centro Socio Sanitario El Carmen, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Not applicable; individual participant data will not be shared.

REFERENCES:
- [Background] Bauer ACM, Andringa G. The Potential of Immersive Virtual Reality for Cognitive Training in Elderly. Gerontology. 2020;66(6):614-623. doi: 10.1159/000509830. Epub 2020 Sep 9. PMID 32906122
- [Background] Liao YY, Chen IH, Lin YJ, Chen Y, Hsu WC. Effects of Virtual Reality-Based Physical and Cognitive Training on Executive Function and Dual-Task Gait Performance in Older Adults With Mild Cognitive Impairment: A Randomized Control Trial. Front Aging Neurosci. 2019 Jul 16;11:162. doi: 10.3389/fnagi.2019.00162. eCollection 2019. PMID 31379553
- [Background] Gomez-Caceres B, Cano-Lopez I, Alino M, Puig-Perez S. Effectiveness of virtual reality-based neuropsychological interventions in improving cognitive functioning in patients with mild cognitive impairment: A systematic review and meta-analysis. Clin Neuropsychol. 2023 Oct;37(7):1337-1370. doi: 10.1080/13854046.2022.2148283. Epub 2022 Nov 23. PMID 36416175
- [Background] Munoz J, Mehrabi S, Li Y, Basharat A, Middleton LE, Cao S, Barnett-Cowan M, Boger J. Immersive Virtual Reality Exergames for Persons Living With Dementia: User-Centered Design Study as a Multistakeholder Team During the COVID-19 Pandemic. JMIR Serious Games. 2022 Jan 19;10(1):e29987. doi: 10.2196/29987. PMID 35044320
- [Background] Papaioannou T, Voinescu A, Petrini K, Stanton Fraser D. Efficacy and Moderators of Virtual Reality for Cognitive Training in People with Dementia and Mild Cognitive Impairment: A Systematic Review and Meta-Analysis. J Alzheimers Dis. 2022;88(4):1341-1370. doi: 10.3233/JAD-210672. PMID 35811514
- [Background] Perra A, Riccardo CL, De Lorenzo V, De Marco E, Di Natale L, Kurotschka PK, Preti A, Carta MG. Fully Immersive Virtual Reality-Based Cognitive Remediation for Adults with Psychosocial Disabilities: A Systematic Scoping Review of Methods Intervention Gaps and Meta-Analysis of Published Effectiveness Studies. Int J Environ Res Public Health. 2023 Jan 14;20(2):1527. doi: 10.3390/ijerph20021527. PMID 36674283
- [Background] Qiu R, Gu Y, Xie C, Wang Y, Sheng Y, Zhu J, Yue Y, Cao J. Virtual reality-based targeted cognitive training program for Chinese older adults: A feasibility study. Geriatr Nurs. 2022 Sep-Oct;47:35-41. doi: 10.1016/j.gerinurse.2022.06.007. Epub 2022 Jul 12. PMID 35839753
- [Background] Zuschnegg J, Schoberer D, Haussl A, Herzog SA, Russegger S, Ploder K, Fellner M, Hofmarcher-Holzhacker MM, Roller-Wirnsberger R, Paletta L, Koini M, Schussler S. Effectiveness of computer-based interventions for community-dwelling people with cognitive decline: a systematic review with meta-analyses. BMC Geriatr. 2023 Apr 12;23(1):229. doi: 10.1186/s12877-023-03941-y. PMID 37041494
- See also: Organización de las Naciones Unidas. (2015). World population ageing. Department of Economic and Social Affairs, Population Division. — https://www.un.org/en/development/desa/population/publications/pdf/ageing/WPA2015_Report.pdf
- See also: Organización Mundial de la Salud. (2023). Demencia, 15 de marzo de 2023. Datos y cifras. — https://www.who.int/es/news-room/fact-sheets/detail/dementia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included two separately recruited pilot groups of patients with mild cognitive impairment (MCI) participating in cognitive stimulation sessions at our outpatient unit. Group 1 (n = 25) was enrolled in Period 1 (Mondays and Wednesdays), and Group 2 (n = 20) in Period 2 (Tuesdays and Thursdays), each after applying inclusion criteria. Each group was independent, with no participant overlap. So the number of participants in Period 2 does not correspond to the number completing Period 1.
Groups:
- Virtual Reality Cognitive Stimulation Program: Participants with MCI undergo 8 VR sessions, using Oculus Quest 2 headsets for immersive cognitive exercises. Activities include a Supermarket Shopping Task for memory, a Payment Task for cognitive flexibility, and a Recipe Sequencing Task for problem-solving. Additionally, 360-degree videos with visuo-verbal stimulation are used to engage attention and episodic memory, monitored by therapists.
  The investigators employ Oculus Quest 2 VR headsets with hand tracking technology to provide a seamless and immersive experience, especially beneficial for participants with Mild Cognitive Impairment (MCI).
  Virtual Reality Cognitive Stimulation Program: Intervention Type: Device Intervention Name: Virtual Reality Cognitive Stimulation Program Description: This program utilizes virtual reality to conduct cognitive stimulation exercises aimed at improving memory, executive functions, and attention in individuals with Mild Cognitive Impairment (MCI). It includes interactive tasks such as virtual shopping, payment simulations, and recipe sequencing, along with 360-degree video sessions for attention and episodic memory training.
  Our pilot for memory stimulation initially targeted 20 participants. However, due to a high number of volunteers, we increased the sample size and organized it into two groups: one with 25 participants and the other with 20. This adjustment ensures robust data collection and analysis.
Period: Pilot Group 1
Arm/Group | Virtual Reality Cognitive Stimulation Program
Started | 25
Completed | 23
Not Completed | 2
Period: Pilot Group 2
Arm/Group | Virtual Reality Cognitive Stimulation Program
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Virtual Reality Cognitive Stimulation Program: Participants with MCI undergo 8 VR sessions, using Oculus Quest 2 headsets for immersive cognitive exercises. Activities include a Supermarket Shopping Task for memory, a Payment Task for cognitive flexibility, and a Recipe Sequencing Task for problem-solving. Additionally, 360-degree videos with visuo-verbal stimulation are used to engage attention and episodic memory, monitored by therapists.
  The investigators employ Oculus Quest 2 VR headsets with hand tracking technology to provide a seamless and immersive experience, especially beneficial for participants with Mild Cognitive Impairment (MCI).
  Virtual Reality Cognitive Stimulation Program: Intervention Type: Device Intervention Name: Virtual Reality Cognitive Stimulation Program Description: This program utilizes virtual reality to conduct cognitive stimulation exercises aimed at improving memory, executive functions, and attention in individuals with Mild Cognitive Impairment (MCI). It includes interactive tasks such as virtual shopping, payment simulations, and recipe sequencing, along with 360-degree video sessions for attention and episodic memory training.
Arm/Group | Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 45
Age, Continuous [Median (Standard Deviation); unit: years] | 75 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 45
Global Cognition State as Measured by the MMSE [Median (Standard Deviation); unit: units on a score 0-30] — MMSE: Mini mental State Examination. Score Range: 0 to 30 points.
  Higher scores means better global cognition function
  units on a score 0-30 | 25.98 (2.02)
Global Cognition State as Measured by the MoCA [Median (Standard Deviation); unit: units on a score 0-30] — MoCA: Montreal Cognitive Assessment.
  Score Range: 0 to 30 points- Higher scores means better global cognition function
  units on a score 0-30 | 17.98 (4.35)
Short Term Verbal Memory as Measured by DST (Forward Span) [Median (Standard Deviation); unit: units on a score 0-9] — DST (forward span): Digit Span Test (forward span). Score Range: 0 to 9points
  - Higher scores indicate better short-term verbal memory. If reporting a score on a scale, please include the unabbreviated scale t
  units on a score 0-9 | 4 (1.07)
Working Memory as Measure by the DST (Backward Span) [Median (Standard Deviation); unit: units on a score 0-9] — DST (backward span): Digit Span Test (backward span). Score Range: 0to 9 points. Higher scores indicate better working memory
  units on a score 0-9 | 3 (0.93)
Visuospatial Attention as Measured by the TMTA [Median (Standard Deviation); unit: seconds] — TMTA: Trial Making Test A. Score Range: Time to complete the test measured in seconds,typically ranging from several seconds to several minutes.
  Lower times (faster completion) indicate better visuospatial attention.
  seconds | 66 (49.42)
Alternating Attention as Measured by the TMTB [Median (Standard Deviation); unit: seconds] — TMTB: Trial Making Test B. Score Range: Time to complete the test measured in seconds, typically ranging from several seconds to several minutes.
  seconds | 202 (425.04)
Processing Speed as Measured by the SDMT [Median (Standard Deviation); unit: number of correct corresponding pairs] — The Symbol Digit Modalities Test (SDMT) measures processing speed, attention, and visual-motor coordination. During the test, participants are required to match abstract symbols with corresponding numbers using a key. The total raw score is calculated as the number of correct symbol-digit pairs completed within a 90-second interval. There is no fixed maximum score, as it varies based on individual performance.
  Higher scores indicate better processing speed and cognitive performance.
  number of correct corresponding pairs | 17 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: Usability of VR Exercises as Measured by an Adapted 8-Item System Usability Scale (SUS)
Description: Adapted 8-Item System Usability Scale (SUS):
  Score Range: 0 to 100 points Interpretation: Higher scores indicate better usability.
Time Frame: immediately post-intervention, within 30 minutes after the last intervention session- 8th session (day 8)
Measure: Mean (Standard Deviation); unit: score on a scale from 0-100
Arm/Group | Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 42
score on a scale from 0-100 | 81.9 (14.9)

2. Primary Outcome: Comfort of VR Headset as Measured by an 8-Item SUS:
Description: Adapted 8-Item VR Headset Comfort Rating:
  Score Range: 0 to 100 points Interpretation: Lower scores indicate better comfort (as most items measure discomfort).
Time Frame: immediately post-intervention, within 30 minutes after the 8th session (day 8)
Measure: Mean (Standard Deviation); unit: score on a scale from 0-100
Arm/Group | Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 42
score on a scale from 0-100 | 86.5 (13.3)

3. Secondary Outcome: Professional´s Usability of VR Exercises as Measured by an Adapted 8-Item SUS:
Description: Scale Title: Professional System Usability Scale (SUS) Score Range: 0 to 100 points Interpretation: Higher scores indicate a professional's perception of better system usability for patient care.
Time Frame: Baseline and immediately post-intervention, within 30 minutes after the 8th session (day 8)
Population: 4 healthcare professionals that have used the VR headsets with patients
Measure: Mean (Standard Deviation); unit: score on a scale from 0-100
Arm/Group | Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 4
score on a scale from 0-100 | 85.2 (10.9)

4. Secondary Outcome: VR Headset Comfort Rating for Professionals as Measured by an Adapted 3-Item SUS:
Description: Scale Title: Professional System Usability Scale (SUS) Score Range: 0 to 100 points Interpretation: Higher scores indicate better comfort and ease of use for the VR headset; lower scores indicate greater discomfort and difficulty with use. This rating is based on a professional assessment of the VR headset's weight, design, and control scheme's impact on patient comfort during use.
Time Frame: immediately post-intervention, within 30 minutes after the 8th session (day 8)
Population: 4 healthcare professionals that have used the VR headset with the patients
Measure: Mean (Standard Deviation); unit: score on a scale from 0-100
Arm/Group | Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 4
score on a scale from 0-100 | 60.4 (22.9)

5. Secondary Outcome: Global Cognition as Measured by the Mini-Mental State Examination (MMSE)
Description: MMSE is a 30-point questionnaire evaluating orientation, attention, recall, language, and visual construction Score Range: 0 to 30 points. Higher scores means better global cognition function
Time Frame: Baseline and immediately post-intervention, within 30 minutes after the 8th session (day 8)
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- Baseline - Virtual Reality Cognitive Stimulation Program; Post-Intervention - Virtual Reality Cognitive Stimulation Program: Participants with MCI undergo 8 VR sessions, using Oculus Quest 2 headsets for immersive cognitive exercises. Activities include a Supermarket Shopping Task for memory, a Payment Task for cognitive flexibility, and a Recipe Sequencing Task for problem-solving. Additionally, 360-degree videos with visuo-verbal stimulation are used to engage attention and episodic memory, monitored by therapists.
  The investigators employ Oculus Quest 2 VR headsets with hand tracking technology to provide a seamless and immersive experience, especially beneficial for participants with Mild Cognitive Impairment (MCI).
  Virtual Reality Cognitive Stimulation Program: Intervention Type: Device Intervention Name: Virtual Reality Cognitive Stimulation Program Description: This program utilizes virtual reality to conduct cognitive stimulation exercises aimed at improving memory, executive functions, and attention in individuals with Mild Cognitive Impairment (MCI). It includes interactive tasks such as virtual shopping, payment simulations, and recipe sequencing, along with 360-degree video sessions for attention and episodic memory training.
Arm/Group | Baseline - Virtual Reality Cognitive Stimulation Program | Post-Intervention - Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 40 | 40
score on a scale | 26 (2.12) | 26.5 (2.3)

6. Secondary Outcome: Global Cognition as Measured by the Montreal Cognitive Assessment (MoCA)
Description: MoCA is a 30-point screening tool for global cognitive function, assessing memory, attention, language, visuospatial skills, and executive function.
  Score Range: 0 to 30 points
  - Higher scores means better global cognition function
Time Frame: Baseline and immediately post-intervention, within 30 minutes after the 8th session (day 8)
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Virtual Reality Cognitive Stimulation Program | Post-Intervention - Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 40 | 40
score on a scale | 19 (4.19) | 20 (4.4)

7. Secondary Outcome: Short-Term Memory as Measured by the Digit Span Test (DST Forward Span)
Description: Forward Digit Span measures verbal short-term memory. Score Range: 0 to 9 points
  - Higher scores indicate better short-term verbal memory.
Time Frame: Baseline and immediately post-intervention, within 30 minutes after the 8th session (day 8)
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Virtual Reality Cognitive Stimulation Program | Post-Intervention - Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 40 | 40
score on a scale | 4.5 (1.1) | 4.5 (0.96)

8. Secondary Outcome: Working Memory as Measured by the Digit Span Test (DST Backward Span)
Description: Backward Digit Span assesses working memory and mental manipulation. Score Range: 0 to 9 points. Higher scores indicate better working memory.
Time Frame: Baseline and immediately post-intervention, within 30 minutes after the 8th session (day 8)
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Virtual Reality Cognitive Stimulation Program | Post-Intervention - Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 40 | 40
score on a scale | 3 (0.97) | 3 (0.77)

9. Secondary Outcome: Visuospatial Attention as Measured by the Trail Making Test Part A (TMT-A)
Description: TMT-A measures visual attention and processing speed. The outcome is time to completion measured in seconds, typically ranging from several seconds to several minutes.
  Lower times (faster completion) indicate better visuospatial attention.
Time Frame: Baseline and immediately post-intervention, within 30 minutes after the 8th session (day 8)
Measure: Median (Standard Deviation); unit: seconds
Arm/Group | Baseline - Virtual Reality Cognitive Stimulation Program | Post-Intervention - Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 40 | 40
seconds | 70.5 (50.4) | 65.5 (38.3)

10. Secondary Outcome: Executive Function as Measured by the Trail Making Test Part B (TMT-B)
Description: TMTB: Trial Making Test B. Score Range: Time to complete the test measured in seconds, typically ranging from several seconds to several minutes.
  Lower times (faster completion) indicate better alternating attention.
Time Frame: Baseline and immediately post-intervention, within 30 minutes after the 8th session (day 8)
Measure: Median (Standard Deviation); unit: seconds
Arm/Group | Baseline - Virtual Reality Cognitive Stimulation Program | Post-Intervention - Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 40 | 40
seconds | 195.5 (421) | 205 (426)

11. Secondary Outcome: Processing Speed as Measured by the Symbol Digit Modalities Test (SDMT)
Description: SDMT: Symbol Digit Modalities Test. The Symbol Digit Modalities Test (SDMT) measures processing speed, attention, and visual-motor coordination. During the test, participants are required to match abstract symbols with corresponding numbers using a key. The total raw score is calculated as the number of correct symbol-digit pairs completed within a 90-second interval. There is no fixed maximum score, as it varies based on individual performance.
  Higher scores indicate better processing speed and cognitive performance.
Time Frame: Baseline and immediately post-intervention, within 30 minutes after the 8th session (day 8)
Measure: Median (Standard Deviation); unit: Number of correct corresponding pairs
Arm/Group | Baseline - Virtual Reality Cognitive Stimulation Program | Post-Intervention - Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 40 | 40
Number of correct corresponding pairs | 17 (9.8) | 18.5 (9.5)

12. Other Pre Specified Outcome: Demographics Variables
Description: Age: numeric
Time Frame: Baseline
Measure: Median (Standard Deviation); unit: years
Arm/Group | Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 40
years | 75.5 (6.19)

13. Other Pre Specified Outcome: Demographics Variables
Description: Gender: 0=female, 1=male, 3=others
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Cognitive Stimulation Program
Number analyzed (Participants) | 40
Participants
  Male | 17
  Female | 23

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 3-month period during the pilot study.
Description: 0
Arm/Group | Virtual Reality Cognitive Stimulation Program
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 2/45
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Virtual Reality Cognitive Stimulation Program (N=45)
Cybersickness (Ear and labyrinth disorders) | 2 (2) — Two participants experienced cybersickness as dizziness. Symptoms resolved in less than 5 minutes after stopping VR. Both participants were willing to continue VR later. One had 3 sessions, and the other had 6 sessions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT06155721/Prot_SAP_ICF_000.pdf